CLINICAL TRIAL: NCT04970290
Title: Face REshaping Effect With Definisse Threads: Clinical and Instrumental Evaluation ( FREE Study)
Brief Title: Clinical and Instrumental Evaluation on Definisse Threads
Acronym: FREE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Relife S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ReGl/20/DTh-Rej/002
Record Dates: First submitted 2021-06-23; First posted 2021-07-21 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2022-04

CONDITIONS: Face
MeSH Terms: conditions — Facies

STUDY DESIGN:
Intervention Model Description: Monocentric, prospective, open label, uncontrolled, post-market clinical investigation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Definisse threads free floating and Definisse threads double needle (Experimental): Definisse™ free floating threads will be used with the Soft Tissue Reshaping-2 (STR-2) Technique, to reposition the tissue of the malar area.
  It is to be used for the face and neck. The thread presents a central area, free of barbs, and two distal areas with barbs. The 12 cm thread will be used in this study.
  Definisse™ double needle thread (12 cm) that is equipped with barbs in the intermediate section, while the side and the central sections are smooth. The thread ends with two straight cut edge needles 10 cm long Definisse™ double needle threads will be used with the Jawline Reshaping (JR) Technique, to reshape the frame of the jawline, lifting the lower face. This is to be used for the face and the neck. The thread ends with two straight cut edge needles The 12 cm thread will be used in this study.
  Interventions: Device: Definisse threads free floating and definisse threads double needle

INTERVENTIONS:
Device: Definisse threads free floating and definisse threads double needle — Definisse threads are two class III medical devices, for evaluate the performance of the reshaping effect of the face at day 30

SUMMARY:
The scope of this clinical trial is to evaluate and confirm thereshaping effect of the face with Definisse Threads double needle and Definisse threads free floating insertion, at day 30. 6 clinical follow up visit will be performed

DETAILED DESCRIPTION:
The scope of this clinical trial is to evaluate and confirm thereshaping effect of the face with Definisse Threads double needle and Definisse threads free floating insertion, at day 30. 6 clinical follow up visit will be performed to evaluate the modification of skin surface characteristics, the reshaping effect of the face, the subject's satisfaction at each visit, the presence/absence of the threads after the implantation and the global pain perception during the implant procedure..

ELIGIBILITY:
Inclusion Criteria:

1. Women, aged between 30 and 60 years (inclusive), looking for aesthetic procedures to improve the aspect of their midface and lower face.
2. Caucasian race.
3. Subjects, as per Investigator's assessment, with the degree of laxity in the middle and lower face belonging to 1-7 classes (inclusive), according to the Facial Laxity Rating Scale.
4. Subjects calm and controlled, according to the Investigator's opinion.
5. Subjects with cooperative attitude, able to comprehend the full nature and the purpose of the investigation, including possible risks, side effects and discomforts and willing to adhere to the study schedule (including attendance to the planned visits) and study prescriptions.
6. Written informed consent release prior to any study-related procedures

Exclusion Criteria:

Absolute exclusion criteria

Subjects presenting one or more of the following absolute exclusion criteria will not be eligible to enter the study.

1. Pregnant and breast-feeding women.
2. Subjects affected by body dysmorphic disorders.
3. Subjects with known allergy/hypersensitivity to threads components and/or lidocaine and/or clarithromycin.
4. Subjects with chronic urticaria.
5. Subjects with Quincke's edema.
6. Subjects with facial plastic surgery within previous 2 years.
7. Subjects with haemostatic or coagulation disorders (haemophilia, haemoglobin pathology, thalassemia major).
8. Subjects with active localized infection (ear, nose, or throat infections, dental abscess, periodontitis), active generalized infection (gastroenteritis, urinary bladder infection) or systemic infection (example: tuberculosis).
9. Subjects with generalized skin conditions or connective tissue disease (prominent scars, keloid, bullous diseases, cutaneous collagenosis, active psoriasis, connective tissue diseases).
10. Subjects with parotid hypertrophy.
11. Immunocompromised, oncological, diabetic subjects or with active Hashimoto's disease.
12. Subjects who underwent dental procedures within previous 2 weeks.
13. Subjects with conditions potentially causing a Koebner response.
14. Subjects with surgical medical treatments previously performed in the implant area or in the surrounding areas within previous 2 months.
15. Subjects with permanent or semi-permanent implants in the area that will be treated.
16. Subjects with active skin infection (impetigo, herpes simplex, massive demodex folliculorum, Pityrosporum, Propionibacterium acnes, viral warts).
17. Obesity.
18. Subjects who are hard smokers (more than 19 cigarettes/day).
19. Any other clinical condition that upon the judgement of the Investigator contraindicates the treatment with threads.

Relative exclusion criteria

Subjects presenting with one or more of the following relative exclusion criteria will be eligible to enter the study on the basis of the Investigator's evaluation.

1. Subjects with severe ptosis.
2. Anxious subjects.
3. Subjects with melasma and post-inflammatory hyperpigmentation.
4. Subjects with non-infectious gastrointestinal conditions like Crohn's disease or ulcerative colitis.
5. Subjects with hypertension, using anti-inflammatory and/or anticoagulant/antiaggregant medications.
6. Subjects who received filler injections or neurotoxin injection within the previous 2 months.
7. Subjects with inflammatory conditions of the skin.
8. Subjects who are mild-moderate smokers.
9. Subjects having menstruation during the day of the treatment.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-11-06 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Volume of midface and lower face with Definisse threads double needle and Definisse threads free floating insertion at day 30 | up to 30 days of treatment
  The primary objective of this clinical investigation is to evaluate the reshaping effect of the face with Definisse™ thread double needle and Definisse™ thread free floating insertion, at Day 30, through 3D photos and 2D photos, through VECTRA®H2

SECONDARY OUTCOMES:
reshaping effect between baseline and T15d, T4m, T8m, T12m. | up to 15 days, 4 months, 8 months and 12 monts of tratment
  To evaluate the reshaping effect of the face with Definisse™ threads between baseline and day 15, 4 months, 8 months, 12 months with GAIS (Global Aesthetic Improvement Scale; 5-item scale, where 1 = exceptional improvement, 2 = very improved, 3 = improved, 4 = unaltered, 5 = worsened.))
To evaluate the modification of skin surface characteristics at 30 days, 4 months, 8 months and 12 monts from baseline | up to 30 days, 4 months, 8 months and 12 monts of tratment
  Modification of skin surface characteristics in terms of wrinkles, pores and texture, that will be evaluated and quantified at day 30d, 4 months, 8 months, 12 months from baseline through ANTERA 3D.
to evaluate the subject's satisfaction at each visit (1 day, 15 days, 30 days, 4 months, 8 months and 12 monts) | up to 1 day, 15 days, 30 days, 4 months, 8 monts and 12 months of treatment
  Subject's satisfaction self-assessment on the reshaping effect according to the Global Aesthetic Improvement Scale (GAIS: 5-item scale, where 1 = exceptional improvement, 2 = very improved, 3 = improved, 4 = unaltered, 5 = worsened.) at each visit (1 day, 15 days, 30 days, 4 months, 8 months and 12 monts).
To assess the clinical evaluation of reshaping effect of the total, middle and lower face comparing baseline to T15d, T30d, T4m, T8m, T12m by the non-treating investigators | up to 15 days, 30 days, 4 months,8 months, 12 months of treatment
  Aesthetic changes of the total, middle and lower face according to the Global Aesthetic Improvement Scale (GAIS: 5-item scale, where 1 = exceptional improvement, 2 = very improved, 3 = improved, 4 = unaltered, 5 = worsened) by the non-treating investigators (one plastic surgeon and one dermatologist) as clinical evaluation of reshaping effect, comparing baseline to T15d, T30d, T4m, T8m, T12m, by evaluating the 2D photos collected by VECTRA®H2
To evaluate the presence/absence of the threads after the implantation at T30d, T4m, T8m, T12m | up to 30 days, 4 months, 8 months, 12 months of treatment
  Presence/absence of the thread in the implant area after 30 days, 4 months, 8 months and 12 monts from the treatment with an ultrasound evaluation.
To evaluate the global pain perception during the implant procedure at T1d and T15d. | up to 1 and 15 days of treatment
  Global pain perception during the implant procedure at 1 day and at the first follow-up visit (15 days) by a numeric pain scale (NRS: from "0" (No pain) to "10" (worst possible pain)).
To evaluate the subject's self-esteem at each visit (1 day, 15 days, 30 days, 4 months, 8 months and 12 monts) T30d, T4m, T8m, T12m). | up to 1 day, 15 ddays, 30 days, 4 months, 8 month, 12 months of treatment
  Subject's self-esteem by the Rosenberg Self-Esteem Scale at each visit ( This scale is a widely used self-report instrument for evaluating individual self-esteem. The scale ranges from 0 to 30. Scores between 15 and 25 are within normal range; scores below 15 suggest low self-esteem.)(1 day, 15 days, 30 days, 4 months, 8 months and 12 monts)

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Fundarò, Principal Investigator — MULTIMED poliambulatorio and day surgery
Locations (1):
- MULTIMED poliambulatorio and day surgery, Bologna, Italia, Italy

IPD SHARING:
Plan to Share IPD: No